CLINICAL TRIAL: NCT02675907
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Evaluation of the Efficacy and Safety of N1539 Following Bunionectomy
Brief Title: Evaluation of N1539 Following Bunionectomy Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baudax Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REC-15-016
Record Dates: First submitted 2016-02-01; First posted 2016-02-05 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Pain, Post-operative
Keywords: Bunion; Bunionectomy; Pain; Analgesia; N1539; Phase 3
MeSH Terms: conditions — Pain, Postoperative; Bunion; Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- N1539 30mg (Experimental): N1539 (Intravenous meloxicam) 30mg every 24 hours for up to 3 doses.
  Interventions: Drug: N1539
- IV Placebo (Placebo Comparator): IV Placebo every 24 hours for up to 3 doses.
  Interventions: Drug: Intravenous Placebo

INTERVENTIONS:
Drug: N1539
  Other Names: Intravenous meloxicam
  Arms: N1539 30mg
Drug: Intravenous Placebo
  Arms: IV Placebo

SUMMARY:
The primary objective of this study is to evaluate the analgesic efficacy of N1539 in subjects with acute moderate to severe pain following unilateral bunionectomy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily provide written informed consent.
* Male or female between 18 and 75 years of age, inclusive.
* Be scheduled to undergo a primary unilateral first metatarsal bunionectomy repair
* Be American Society of Anesthesiology (ASA) physical class 1 or 2.
* Female subject are eligible only if all the following apply:

  * Not pregnant;
  * Not lactating;
  * Not planning to become pregnant during the study;
  * Commit to the use of an acceptable form of birth control for the duration of the study.
* Have a body mass index ≤35 kg/m2
* Be able to understand the study procedures, comply with all study procedures, and agree to participate in the study program.

Exclusion Criteria:

* Have a known allergy to meloxicam or any excipient of N1539, D5W, aspirin, other non-steroidal anti-inflammatory drugs (NSAIDs) or to any peri- or postoperative medications used in this study.
* Have a clinically significant abnormal clinical laboratory test value.
* Have history of or positive test results for HIV, or hepatitis B or C.
* Have a history or clinical manifestations of significant renal, hepatic, cardiovascular, metabolic, neurologic, psychiatric, or other condition that would preclude participation in the study.
* Have a history of myocardial infarction or coronary artery bypass graft surgery within the preceding 12 months
* Have a history of migraine or frequent headaches, seizures, or are currently taking anticonvulsants.
* Have active or recent (within 6 months) gastrointestinal ulceration or bleeding.
* Have a known bleeding disorder or be taking agents affecting coagulation
* Have another painful physical condition that may confound the assessments of post operative pain.
* Have evidence of a clinically significant 12 lead ECG abnormality.
* Have a history of alcohol abuse (regularly drinks > 4 units of alcohol per day; 8 oz. beer, 3 oz. wine, 1 oz. spirits) within the past 5 years or a history of prescription/illicit drug abuse.
* Have positive results on the urine drug screen or alcohol breath test indicative of illicit drug or alcohol abuse.
* Have been receiving or have received chronic opioid therapy defined as greater than 15 morphine equivalents units per day for greater than 3 out of 7 days per week over a one-month period within 12 months of surgery.
* Use concurrent therapy that could interfere with the evaluation of efficacy or safety, such as any drugs which in the investigator's opinion may exert significant analgesic properties or act synergistically with N1539.
* Unable to discontinue medications, that have not been at a stable dose for at least 14 days prior to the scheduled bunionectomy procedure, within 5 half lives of the specific prior medication (or, if half life is not known, within 48 hours) before dosing with study medication.
* Have utilized corticosteroids, either systemically or by intra-articular injection, within 6 weeks prior to the surgical procedure.
* Have received any investigational product within 30 days before dosing with study medication.
* Be receiving warfarin, lithium, or a combination of furosemide with either an angiotensin converting enzyme inhibitor or an angiotensin receptor blocker
* Be currently receiving treatment with oral meloxicam (Mobic®) within 7 days prior to surgery
* Have previously received N1539 in clinical trials, or had major surgery in the last 3 months that would interfere with study outcomes or increase the risk of study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Trovare Clinical Research, Bakersfield, California
  - Lotus Clinical Research, Pasadena, California
  - Chesapeake Research Group, Pasadena, Maryland
  - Endeavor Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Viscusi ER, Gan TJ, Bergese S, Singla N, Mack RJ, McCallum SW, Du W, Hobson S. Intravenous meloxicam for the treatment of moderate to severe acute pain: a pooled analysis of safety and opioid-reducing effects. Reg Anesth Pain Med. 2019 Mar;44(3):360-368. doi: 10.1136/rapm-2018-100184. Epub 2019 Feb 7. PMID 30737315

RESULTS

PARTICIPANT FLOW:
Groups:
- N1539 30 mg: N1539 (Intravenous meloxicam) 30 mg every 24 hours for up to 3 doses.
  N1539
- IV Placebo: IV Placebo every 24 hours for up to 3 doses.
  Intravenous Placebo
Period: Treatment Phase (48 Hours Post-Dose 1)
Arm/Group | N1539 30 mg | IV Placebo
Started | 100 | 101
Completed | 95 | 96
Not Completed | 5 | 5
Not completed — Lack of Efficacy | 4 | 4
Not completed — Withdrawal by Subject | 1 | 1
Period: Study Overall
Arm/Group | N1539 30 mg | IV Placebo
Started | 100 | 101
Completed | 97 | 97
Not Completed | 3 | 4
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N1539 30 mg | IV Placebo | Total
Number analyzed (Participants) | 100 | 101 | 201
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 92 | 92 | 184
  >=65 years | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (12.79) | 48.4 (12.17) | 47.6 (12.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 87 | 171
  Male | 16 | 14 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 36 | 64
  Not Hispanic or Latino | 72 | 65 | 137
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 32 | 26 | 58
  White | 61 | 68 | 129
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100 | 101 | 201
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.9 (4.80) | 28.3 (4.02) | 27.6 (4.46)
Time from End of Surgery to First Dose [Mean (Standard Deviation); unit: hours] | 0.514 (0.2397) | 0.485 (0.2001) | 0.500 (0.2206)
Baseline Pain Intensity [Mean (Standard Deviation); unit: units on a scale] — Pain Intensity was assessed using the 11-point Numeric Pain Rating Scale (NPRS; 0-10) with the baseline assessment being the NPRS score collection prior to the first study dose.
  units on a scale | 6.7 (1.90) | 7.0 (1.82) | 6.8 (1.86)

OUTCOME MEASURES:

1. Primary Outcome: Summed Pain Intensity Difference Over the First 48 Hours (SPID48)
Description: Pain intensity was recorded using a Numeric Pain Rating Scale (Range 0-10) where 0 equates to no pain (better), and 10 equates to the worst pain imaginable (worse). Pain intensity scores were to be recorded at the following time points: 0.25, 0.5, 0.75, 1, and 2 hours post Dose 1. Thereafter pain assessments were to be recorded every 2 hours until 48 hours post Dose 1. Pain intensity differences from baseline at each time point were calculated and a time weighted summed pain intensity difference (SPID) was then calculated. Time weighted SPID calculations were computed by multiplying a weight factor to each score prior to summation. The weight factor at each time point was the time elapsed since the previous observation. A smaller SPID value (i.e. more negative) was better.
Time Frame: 48 Hours
Population: Intent-to-Treat (ITT) population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | N1539 30 mg | IV Placebo
Number analyzed (Participants) | 100 | 101
units on a scale | -6956.0 (521.69) | -4829.3 (519.56)
Statistical Analysis 1: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p = 0.0034, t-test, 2 sided

2. Secondary Outcome: Summed Pain Intensity Difference (SPID) at Other Intervals
Description: as for outcome 1
Time Frame: 48 Hours
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | N1539 30 mg | IV Placebo
Number analyzed (Participants) | 100 | 101
units on a scale
  SPID6 (Hour 0-6) | -510.78 (66.22) | -288.33 (65.95)
  SPID12 (Hour 0-12) | -957.83 (123.30) | -480.15 (122.80)
  SPID24 (Hour 0-24) | -2071.0 (247.01) | -1167.9 (246.00)
  SPID12-48 (Hour 12-48) | -5998.2 (439.21) | -4349.1 (437.42)
  SPID24-48 (Hour 24-48) | -4885.1 (313.60) | -3661.4 (312.32)
Statistical Analysis 1: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p < 0.05, t-test, 2 sided — Row 1 (SPID6)
Statistical Analysis 2: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p < 0.01, t-test, 2 sided — Row 2 (SPID12)
Statistical Analysis 3: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p < 0.01, t-test, 2 sided — Row 3 (SPID24)
Statistical Analysis 4: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p < 0.01, t-test, 2 sided — Row 4 (SPID12-48)
Statistical Analysis 5: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p < 0.01, t-test, 2 sided — Row 5 (SPID24-48)

3. Secondary Outcome: Time to First Dose of Rescue Analgesia
Description: Rescue analgesia (oral oxycodone 5 mg) was available to subjects with inadequately controlled pain upon request. Time to first rescue was calculated as the elapsed time from administration of Dose 1 to the administration of the first dose of rescue analgesia.
Time Frame: 48 Hours
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | N1539 30 mg | IV Placebo
Number analyzed (Participants) | 100 | 101
hours | 1.99 [1.53 to 4.12] | 2.09 [1.15 to 3.31]
Statistical Analysis 1: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p = 0.0076, Log Rank

4. Secondary Outcome: Number of Subjects Utilizing Rescue Analgesia
Description: Rescue analgesia (oral oxycodone 5 mg) was available to subjects with inadequately controlled pain upon request.
Time Frame: 48 Hours
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | N1539 30 mg | IV Placebo
Number analyzed (Participants) | 100 | 101
Participants
  Hour 0-24 | 83 | 99
  Hour 24-48 | 48 | 71
  Hour 0-48 | 83 | 99
Statistical Analysis 1: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Row 1 (Hour 0-24)
Statistical Analysis 2: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p < 0.01, Cochran-Mantel-Haenszel — Row 2 (Hour 24-48)
Statistical Analysis 3: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p < 0.01, Cochran-Mantel-Haenszel — Row 3 (Hour 0-48)

5. Secondary Outcome: Number of Doses of Rescue Analgesia Utilized Per Subject
Description: Rescue analgesia (oral oxycodone 5 mg) was available to subjects with inadequately controlled pain upon request.
Time Frame: 48 Hours
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: doses of rescue analgesia
Arm/Group | N1539 30 mg | IV Placebo
Number analyzed (Participants) | 100 | 101
doses of rescue analgesia
  Hour 0-24 | 3.97 (0.26) | 5.06 (0.26)
  Hour 24-48 | 1.63 (0.25) | 2.51 (0.25)
  Hour 0-48 | 5.45 (0.46) | 7.49 (0.46)
Statistical Analysis 1: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p < 0.05, ANCOVA — Row 1 (Hour 0-24); P-values were derived from ANCOVA models with fixed effects of treatment, baseline PI score, and investigational site
Statistical Analysis 2: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p < 0.05, ANCOVA — Row 2 (Hour 24-48); P-values were derived from ANCOVA models with fixed effects of treatment, baseline PI score, and investigational site
Statistical Analysis 3: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p < 0.05, ANCOVA — Row 3 (Hour 0-48); P-values were derived from ANCOVA models with fixed effects of treatment, baseline PI score, and investigational site

6. Secondary Outcome: Time to Perceptible Pain Relief (TTPPR)
Description: Time to perceptible and meaningful pain relief was measured using the double stopwatch method. For each randomized subject, two stopwatches were started immediately after administration of the first study dose (Hour 0). The subject was to stop the first watch when they first perceived pain relief to occur (time to perceptible relief). Once the first watch was stopped, the second stopwatch was given to the subject with the instructions to stop the watch when they first experienced meaningful pain relief (time to meaningful relief).
Time Frame: 12 Hours
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | N1539 30 mg | IV Placebo
Number analyzed (Participants) | 100 | 101
hours | 0.52 [0.35 to 0.74] | 1.59 [0.48 to 2.00]
Statistical Analysis 1: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p = 0.1228, Log Rank

7. Secondary Outcome: Time to Meaningful Pain Relief (TTMPR)
Description: as for outcome 6
Time Frame: 12 Hours
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | N1539 30 mg | IV Placebo
Number analyzed (Participants) | 100 | 101
hours | 2.16 [1.00 to 12.01] | 3.19 [2.39 to 4.82]
Statistical Analysis 1: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p = 0.1048, Log Rank

8. Secondary Outcome: Subjects With ≥ 30% Improvement in Pain From Baseline to Hour 6
Description: Percent improvement in pain is the cumulative pain intensity percent reduction from baseline over the defined interval (6 or 24 hours), calculated as SPID for the defined interval (SPID6 or SPID24) divided by the baseline pain intensity (BaselinePI) extrapolated across that interval. Example: % Improvement through Hour 6 = 100 * SPID6 / (BaselinePI * 6 * 60), and SPID6 < 0 as an indication for improvement.
Time Frame: 6 Hours
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | N1539 30 mg | IV Placebo
Number analyzed (Participants) | 100 | 101
Participants | 32 | 20
Statistical Analysis 1: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p = 0.0451, Cochran-Mantel-Haenszel

9. Secondary Outcome: Subjects With ≥ 30% Improvement in Pain From Baseline to Hour 24
Description: Percent improvement in pain is the cumulative pain intensity percent reduction from baseline over the defined interval (6 or 24 hours), calculated as SPID for the defined interval (SPID6 or SPID24) divided by the baseline pain intensity (BaselinePI) extrapolated across that interval. Example: % Improvement through Hour 24 = 100 * SPID24 / (BaselinePI * 24 * 60), and SPID24 < 0 as an indication for improvement.
Time Frame: 24 Hours
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | N1539 30 mg | IV Placebo
Number analyzed (Participants) | 100 | 101
Participants | 37 | 21
Statistical Analysis 1: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p = 0.0107, Cochran-Mantel-Haenszel

10. Secondary Outcome: Subjects With ≥ 50% Improvement in Pain From Baseline to Hour 6
Description: as for outcome 8
Time Frame: 6 Hours
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | N1539 30 mg | IV Placebo
Number analyzed (Participants) | 100 | 101
Participants | 16 | 8
Statistical Analysis 1: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p = 0.0781, Cochran-Mantel-Haenszel

11. Secondary Outcome: Subjects With ≥ 50% Improvement in Pain From Baseline to Hour 24
Description: as for outcome 9
Time Frame: 24 Hours
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | N1539 30 mg | IV Placebo
Number analyzed (Participants) | 100 | 101
Participants | 13 | 5
Statistical Analysis 1: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p = 0.0430, Cochran-Mantel-Haenszel

12. Secondary Outcome: Patient Global Assessment (PGA) of Pain Control at Hour 24
Description: PGA of pain control was evaluated at Hour 24 and Hour 48 with subject reported degree of pain control over the preceding interval according to a 5 point scale (0-4) with categories of 0-poor, 1-fair, 2-good, 3-very good, or 4-excellent.
Time Frame: 24 Hours
Measure: Count of Participants; unit: Participants
Arm/Group | N1539 30 mg | IV Placebo
Number analyzed (Participants) | 95 | 97
Participants
  0 - Poor | 17 | 29
  1 - Fair | 23 | 26
  2 - Good | 28 | 26
  3 - Very Good | 17 | 13
  4 - Excellent | 10 | 3
Statistical Analysis 1: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p = 0.1070, Cochran-Mantel-Haenszel; P-value was derived from comparisons between N1539 and Placebo via General Association of CMH Test controlling for investigational site

13. Secondary Outcome: Patient Global Assessment (PGA) of Pain Control at Hour 48
Description: as for outcome 12
Time Frame: 48 Hours
Measure: Count of Participants; unit: Participants
Arm/Group | N1539 30 mg | IV Placebo
Number analyzed (Participants) | 95 | 96
Participants
  0 - Poor | 7 | 15
  1 - Fair | 8 | 18
  2 - Good | 26 | 25
  3 - Very Good | 30 | 30
  4 - Excellent | 24 | 8
Statistical Analysis 1: Comparison: N1539 30 mg vs IV Placebo; Test type: Superiority; p = 0.0046, Cochran-Mantel-Haenszel; [statistical method as in outcome 12, analysis 1]

ADVERSE EVENTS:
Time Frame: AEs collected from time of first dose through last followup (30 days)
Arm/Group | N1539 30 mg | IV Placebo
All-Cause Mortality (participants affected / at risk) | 0/100 | 1/101
Serious Adverse Events (participants affected / at risk) | 0/100 | 2/101
Other Adverse Events (participants affected / at risk) | 44/100 | 54/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N1539 30 mg (N=100) | IV Placebo (N=101)
Sudden death (General disorders) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N1539 30 mg (N=100) | IV Placebo (N=101)
Nausea (Gastrointestinal disorders) | 20 (30) | 26 (31)
Constipation (Gastrointestinal disorders) | 4 (4) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 9 (11)
Injection site erythema (General disorders) | 0 (0) | 2 (2)
Injection site pain (General disorders) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Incision site cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 2 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 7 (8)
Dizziness (Nervous system disorders) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 8 (8) | 12 (14)
Somnolence (Nervous system disorders) | 3 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8) | 3 (3)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Flushing (Vascular disorders) | 3 (4) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Discussion and/or publication of data generated is not permitted without the prior written consent of the sponsor.